CLINICAL TRIAL: NCT06102447
Title: Efficacy and Safety of Netupitant and Palonosetron Hydrochloride Capsules in Preventing Nausea and Vomiting Induced by Radiochemotherapy in Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Yangkun Luo, Study Director, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCHEC-02-2023-076
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Drug: Netopitam Palonosetron capsules and dexamethasone

INTERVENTIONS:
Drug: Netopitam Palonosetron capsules and dexamethasone — On the first and third days, they took Netopitam Palonosetron capsules and dexamethasone to reduce the incidence of acute vomiting.

SUMMARY:
The enrolled head and neck squamous cell carcinoma patients in this study received high-dose multiday chemotherapy with cisplatin and synchronous radiation therapy, which had a high risk of nausea and vomiting. On the first and third days, they took Netopitam Palonosetron capsules and dexamethasone to reduce the incidence of acute vomiting. The aim of this study is to evaluate the antiemetic effect of Netopitam Palonosetron capsules and to explore the effectiveness of using Netopitam Palonosetron capsules again for antiemetic treatment during the study period when breakthrough vomiting occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18-75 years old;
2. Head and neck tumors confirmed by histology or cytology (including oral cancer, oropharyngeal cancer, hypopharyngeal cancer, and laryngeal cancer);
3. Receive radical synchronous radiotherapy and chemotherapy;
4. The Eastern Oncology Collaborative Group (ECOG) physical fitness score of the subjects was ≤ 2 points;
5. Adequate organ and bone marrow function;
6. The expected life is at least 12 weeks;
7. Pregnant or fertile patients (male or female) use reliable contraceptive measures;
8. When screening female patients with potential pregnancy, the pregnancy test must be negative;
9. The subjects voluntarily and strictly comply with the requirements of the research protocol and sign a written informed consent form.

Exclusion Criteria:

1. Recurrent and metastatic head and neck tumors;
2. Previously underwent tumor resection surgery for treatment;
3. Patients with platinum drug intolerance;
4. Receiving any known or potential antiemetic medication within 24 hours prior to the first day, or experiencing symptoms of vomiting, retching, or mild nausea within 24 hours prior to the first day;
5. Take NK1（neurokinin-1） receptor antagonists or any study medication within 4 weeks before the start of the experiment;
6. Use CYP3A4 inducer within 4 weeks before chemotherapy, and use CYP3A4 substrate or strong or moderate CYP3A4 inhibitor within 1 week;
7. Serious cardiovascular, pulmonary, diabetes, mental and other diseases;
8. Pregnant or lactating women, patients with fertility who are unwilling or unable to take effective contraceptive measures;
9. Drug and/or alcohol abuse;
10. Hypocalcemia or any other condition that may cause vomiting;
11. There are significant factors that affect the absorption of oral medication, such as chronic diarrhea and intestinal obstruction;
12. The subject has allergic reactions to Netopitam Palonosetron capsules or any of their excipients;
13. Within 30 days prior to the baseline visit, the subject participated in another clinical study and used any exploratory drugs or devices; Allow participation in observational research;
14. The researcher determines other situations that may affect the progress of clinical research and the determination of research results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The complete response rate during synchronous radiotherapy and chemotherapy (defined as no vomiting episodes and no emergency medication). | 1 month

SECONDARY OUTCOMES:
No significant nausea rate during synchronous radiotherapy and chemotherapy | 1 month
Nausea free rate during synchronous radiotherapy and chemotherapy | 1 month
No vomiting rate during synchronous radiotherapy and chemotherapy | 1 month
The rate of non emergency medication during synchronous radiotherapy and chemotherapy | 1 month
The prevalence and severity of oral/oropharyngeal mucositis during synchronous radiotherapy and chemotherapy | 1 month
Successful rescue rate of breakthrough vomiting: (defined as no vomiting within 48 hours) | 1 month
Evaluate the impact of medication on patients' daily activities of life (evaluated based on the nausea and vomiting questionnaire FLIE) | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China